CLINICAL TRIAL: NCT05473338
Title: Comparison of Gut Microbial Composition and Function in CRPS Patients vs. Healthy Individuals
Brief Title: Complex Regional Pain Syndrome (CRPS) and the Gut-bacteria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Louise and Alan Edwards Foundation (Unknown); Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Yoram Shir, Director, the Alan Edwards Pain Management Unit, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: CRPS-MB 2021-6735
Record Dates: First submitted 2022-04-12; First posted 2022-07-25 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: CRPS
MeSH Terms: interventions — Defecation; Blood Specimen Collection; Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRPS (Complex Regional Pain Syndrome): Participants with CRPS (Complex Regional Pain Syndrome))
  Interventions: Diagnostic Test: Stool and blood samples; Other: Physical examination; Other: Questionnaires
- Healthy: Healthy individuals
  Interventions: Diagnostic Test: Stool and blood samples; Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Stool and blood samples — fecal microbiome and metabolomics, as well as metabolites in plasma
Other: Physical examination — physical examination performed by a physician to confirm CRPS diagnosis and assess patient's eligibility to participate in the study. The exam will include skin temperature measured using a laser/infrared skin thermometry.
  Groups: CRPS (Complex Regional Pain Syndrome)
Other: Questionnaires — Questionnaires measuring pain level, sleep, mood and diet parameters.

SUMMARY:
The purpose of this study is to investigate, for the first time, whether gut bacteria composition and function of patients with CRPS differ from those of healthy adults. Samples of stool, urine and blood will be collected from patients with CRPS and from healthy adults. The type and function of bacteria of CRPS patients will be analyzed and compared to those of healthy adults to test if potential differences could explain the mechanism/s involved with the development of CRPS.

ELIGIBILITY:
Inclusion criteria:

1. Women and men over the age of 18, diagnosed with CRPS of the upper or lower limb according to the Clinical Budapest Criteria, with a duration of 6 months and over (for the 1st study group).
2. Healthy women and men over the age of 18, who share a household with a CRPS patients participating in the study (for the 1st control group).
3. Healthy women and men over the age of 18 (for the 2nd control group).
4. Be able to read and write in either French, English or Hebrew.

Exclusion criteria:

1. Any major illness (eg. malignancy, active inflammatory disease, metabolic disease, etc.)
2. Pregnancy
3. Chronic pain conditions (other than CRPS in the patients group)
4. Acute illness of any type in the preceding 1 month
5. Use of systemic antibiotics in the preceding 1 month
6. Change in any other regularly taken medications in the past 1 month
7. Substantial dietary / gastrointestinal alterations in the past 1 month.

The inclusion/exclusion criteria were set to reduce the risk of confounding factors that could affect gut microbiota composition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women and men with CRPS and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | 1 day
  Assessment of genomic composition of the gut bacteria by differential abundance analysis will be performed using 16S rRNA (Genome-Quebec)
Presence of stool microbiota-related metabolites affecting host physiology | 1 day
  Concentration of bile acids and short-chain-fatty-acids through Metabolomics analysis (Metabolon, USA).

SECONDARY OUTCOMES:
Short-form health-questionnaire (SF12) score | 1 day
  A 12-item measure of health-related quality of life, validated in a variety of population groups
Brief Pain Inventory (BPI) score | 1 day
  A 12-item questionnaire evaluating function level and disability among pain patients
Patient Health Questionnaire (PHQ-9) score | 1 day
  A 9 item inventory rated on a 4 point Likert-type scale used for screening for depression and anxiety
Pittsburg Sleep Quality Index (PSQI) scores | 1 day
  A standardized self-administered questionnaire for the assessment of subjective sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Shir, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Alan Edwards Pain Management Unit - Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birklein F, Ajit SK, Goebel A, Perez RSGM, Sommer C. Complex regional pain syndrome - phenotypic characteristics and potential biomarkers. Nat Rev Neurol. 2018 May;14(5):272-284. doi: 10.1038/nrneurol.2018.20. Epub 2018 Mar 16. PMID 29545626
- [Background] Birklein F, O'Neill D, Schlereth T. Complex regional pain syndrome: An optimistic perspective. Neurology. 2015 Jan 6;84(1):89-96. doi: 10.1212/WNL.0000000000001095. Epub 2014 Dec 3. PMID 25471395
- [Background] Harden RN, Bruehl S, Stanton-Hicks M, Wilson PR. Proposed new diagnostic criteria for complex regional pain syndrome. Pain Med. 2007 May-Jun;8(4):326-31. doi: 10.1111/j.1526-4637.2006.00169.x. PMID 17610454
- [Background] Minerbi A, Gonzalez E, Brereton NJB, Anjarkouchian A, Dewar K, Fitzcharles MA, Chevalier S, Shir Y. Altered microbiome composition in individuals with fibromyalgia. Pain. 2019 Nov;160(11):2589-2602. doi: 10.1097/j.pain.0000000000001640. PMID 31219947